CLINICAL TRIAL: NCT07224334
Title: Alpha to Beta Cell Communication in Health and Disease
Brief Title: Role of Alpha-to-beta Cell Communication to Adapt Insulin Secretion to Insulin Resistance.
Acronym: UPGRADE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David D'Alessio, M.D. (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, David D'Alessio, M.D., Professor of Medicine Duke University, Director Division of Endocrinology, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00116631; R01DK142423 (NIH)
Record Dates: First submitted 2025-10-29; First posted 2025-11-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Diabetes (DM)
Keywords: insulin secretion; insulin sensitivity; GLP-1; alpha- to beta-cell communication
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Each subject will have paired, single day experiments performed within 4-5 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Aim 2A: Glucose-stimulated insulin secretion with and without GLP-1 receptor blockade (Placebo Comparator): Aim 2A: Each subject will have a 5 hr experiment with sequential hyperglycemic clamps separated by a 90-minute washout. Blood glucose will be increased with an intravenous (IV) infusion of 20% dextrose and maintained stable at a level of 2.5-3.0 mM above fasting glucose for 90 minutes. Following the washout, a second, identical hyperglycemic clamp will be performed. Subjects will receive either saline or exendin-9 (600 pmol/kg/min) during the clamps; in 10 subjects the saline/clamp will be first and in 10 subjects the exendin-9/clamp will be first; the orders will be assigned randomly.
  Intervention: The interventions here are the experimental hyperglycemia with and without exendin-9
  Interventions: Drug: Exendin-9 is a 30 amino acid peptide that is an established competitive antagonist of the GLP-1 receptor. Subjects will receive exendin-9 by intravenous infusion at a rate of 600 pmol/kg/min
- Glucose stimulated insulin secretion with or without GLP-1 receptor blockade and insulin resistance (Active Comparator): Aim 2A: Subjects will be treated with 6 mg dexamethasone once daily for 7 days to induce insulin resistance before repeating the 5 hr glucose clamp study. The infusion of glucose with saline and exendin-9 will be performed identically to the first study.
  Intervention: The intervention in this arm is the induction of insulin resistance with dexamethasone treatment.
  Interventions: Drug: Exendin-9 is a 30 amino acid peptide that is an established competitive antagonist of the GLP-1 receptor. Subjects will receive exendin-9 by intravenous infusion at a rate of 600 pmol/kg/min
- Aim 2B: Glucose stimulated insulin secretion and insulin sensitivity (Placebo Comparator): Aim 2B: Each subject will have a 3-hour experiment with a 90-minute hyperglycemic clamp at a level of 2.5-3.0 mM above fasting glucose followed by a 60 minute hyperinsulinemic (80 units/meter2 Body Surface Area/minute), euglycemic clamp.
  Interventions: Drug: Dexamethasone
- Aim 2B: Glucose stimulated insulin secretion with GLP-1 receptor blockade and insulin sensitivity (Active Comparator): Aim 2B: Subjects will have an identical hyperglycemic clamp but with infusion of exendin-9 (600 pmol/kg/min). Exendin-9 infusion will be stopped before the following hyperinsulinemic clamp that will be conducted identically to the control arm. Allocation of subjects in Aim 2B to the study with and without exendin-9 will be randomized.
  Intervention: The intervention in this study is the administration of exendin-9 during experimental hyperglycemia.
  Interventions: Drug: Exendin-9 is a 30 amino acid peptide that is an established competitive antagonist of the GLP-1 receptor. Subjects will receive exendin-9 by intravenous infusion at a rate of 600 pmol/kg/min

INTERVENTIONS:
Drug: Exendin-9 is a 30 amino acid peptide that is an established competitive antagonist of the GLP-1 receptor. Subjects will receive exendin-9 by intravenous infusion at a rate of 600 pmol/kg/min — Subjects in Aim 2A will receive exendin-9 on both experimental days and dexamethasone for one week before their second experimental day.
  Subjects in Aim 2B will receive exendin-9 on one of their two experimental days.
  Arms: Aim 2A: Glucose-stimulated insulin secretion with and without GLP-1 receptor blockade; Aim 2B: Glucose stimulated insulin secretion with GLP-1 receptor blockade and insulin sensitivity; Glucose stimulated insulin secretion with or without GLP-1 receptor blockade and insulin resistance
Drug: Dexamethasone — Dexamethasone 6 mg daily
  Arms: Aim 2B: Glucose stimulated insulin secretion and insulin sensitivity

SUMMARY:
Glucagon secretion from α-cells has long been viewed as primarily a counterregulatory mechanism - e.g. an agent with a role to prevent blood sugar from decreasing to levels that compromise function. Our group, along with other researchers, have begun to identify a much more complex role for α-cells, raising questions about when and how glucagon may influence blood glucose levels. This proposal looks to detail proglucagon peptide secretion from α-cells and the impact this has on β-cell function and glucose tolerance, in preclinical studies of human islets and translational studies in human subjects.

This protocol registration describes Aim 2 from this NIH grant which involves 2 study populations and separate protocols but addresses a common question. Aim 3 in the grant is focused on a separate hypothesis and will be conducted and published separately from Aim 2.

DETAILED DESCRIPTION:
Subjects will undergo screening for medical history, medication usage, and blood work; those who qualify will be offered participation. Study participation will last approximately 4-5 weeks depending on appointment availability.

Aim 2A: Each participant will have two 5-hour hyperglycemic clamp procedures to test the effect of fasting glucagon-like peptide 1 (GLP-1) action before and after experimental insulin resistance. The effect of endogenous proglucagon peptides (glucagon and GLP-1) to stimulate insulin secretion will be determined by blockade of the GLP-1 receptor with the antagonist exendin-9 (Ex-9) during glucose infusions. Insulin secretion experiments will be repeated before and after induction of insulin resistance. To induce insulin resistance, subjects will take dexamethasone, a synthetic glucocorticoid that has been shown in published studies and in a pilot study by our group to reduce insulin sensitivity by ~30%.

Aim 2B: This study will recruit non-diabetic subjects with obesity. They will be studied on two occasions using a 4.5-hour procedure with a hyperglycemic clamp to measure insulin secretion, followed by a hyperinsulinemic, euglycemic clamp to measure insulin sensitivity. This procedure will be done 2 times, once with saline infused during hyperglycemia as a control, and once with exendin-9 given during hyperglycemia to determine the role of GLP-1 receptor action.

ELIGIBILITY:
Aim 2A: Inclusion Criteria:

* Age 18-45
* Body Mass Index (BMI) < 27.0
* Fasting plasma glucose of ≤ 95 mg/dL or HbA1c value ≤ 5.8% as measured at screening visit

Exclusion Criteria:

* Active medical disease: e.g. active infectious, inflammatory, neurodegenerative or mental health disorders
* Personal history of diabetes or pancreatitis
* Personal history of cardiac, gastrointestinal, renal or liver disease
* Immediate family history of diabetes
* Renal insufficiency (eGFR < 60 mL/kg/min)
* Anemia (hematocrit < 34%) as measured at screening visit
* Pregnant females
* Poor vein access
* Consumption of daily medications that alter glucose metabolism of GI function (glucocorticoids, psychotropics, narcotics, metoclopramide)
* Apparent sensitivity to the study peptide as determined by the skin test

Aim 2B: Inclusion Criteria:

* Age 35-60
* Body Mass Index (BMI) ≥ 27.0
* Fasting plasma glucose of < 126 mg/dL or HbA1c value < 6.5% as measured at screening visit

Exclusion Criteria:

* Active medical disease: e.g. active infectious, inflammatory, neurodegenerative or mental health disorders
* Personal history of diabetes or pancreatitis
* Personal history of cardiac, gastrointestinal, renal or liver disease
* Immediate family history of diabetes
* Renal insufficiency (eGFR < 60 mL/kg/min)
* AST and/or ALT levels > 3x the upper limit of the normal range
* Anemia (hematocrit < 34%) as measured at screening visit
* Pregnant females
* Poor vein access
* Consumption of daily medications that alter glucose metabolism of GI function (glucocorticoids, psychotropics, narcotics, metoclopramide)
* Apparent sensitivity to the study peptide as determined by the skin test

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Insulin secretion | Insulin secretion rates will be measured on both days of study in subjects participating in Aims 2A and 2B. Studies will be completed over a period of 4-5 weeks
  Insulin secretion rates will be computed from deconvolution of C-peptide concentrations measured from plasma samples taken during the hyperglycemic clamps.
Insulin secretion with and without exendin-9: Aims 2A and 2B | 4-5 weeks
  Insulin secretion rates derived from deconvolution of C-peptide will be the primary outcome for insulin secretion. This measure will be compared within subjects in Aim 2A with the difference between the saline and exendin-9 clamps on each day used as the measure of fasting GLP-1 receptor mediated insulin secretion. Comparison of GLP-1 receptor mediated insulin secretion between the placebo and dexamethasone studies will be used to determine the effect of insulin resistance.
  Insulin secretion rates will also be compared within subjects in Aim 2B. Here the two different study days, one with saline and one with exendin-9 will be used.

SECONDARY OUTCOMES:
Insulin sensitivity: Aim 2B | Insulin sensitivity will be measured in subjects participating in Aim 2B during the hyperinsulinemic clamp in each of the two days of study. The two experiments will be completed in a 4-5 week period.
  Insulin sensitivity will be measured directly in subjects in Aim 2B during the hyperinsulinemic, euglycemic clamp. The glucose infusion rate necessary to maintain blood glucose a 4-5 mM divided by steady-state plasma insulin will be used as the index of insulin sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: David D'Alessio, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryan AS, Muller DC, Elahi D. Sequential hyperglycemic-euglycemic clamp to assess beta-cell and peripheral tissue: studies in female athletes. J Appl Physiol (1985). 2001 Aug;91(2):872-81. doi: 10.1152/jappl.2001.91.2.872. PMID 11457805
- [Background] Jensen DH, Aaboe K, Henriksen JE, Volund A, Holst JJ, Madsbad S, Krarup T. Steroid-induced insulin resistance and impaired glucose tolerance are both associated with a progressive decline of incretin effect in first-degree relatives of patients with type 2 diabetes. Diabetologia. 2012 May;55(5):1406-16. doi: 10.1007/s00125-012-2459-7. PMID 22286551
- [Background] Salehi M, Vahl TP, D'Alessio DA. Regulation of islet hormone release and gastric emptying by endogenous glucagon-like peptide 1 after glucose ingestion. J Clin Endocrinol Metab. 2008 Dec;93(12):4909-16. doi: 10.1210/jc.2008-0605. Epub 2008 Sep 30. PMID 18827000
- [Background] Gray SM, Goonatilleke E, Emrick MA, Becker JO, Hoofnagle AN, Stefanovski D, He W, Zhang G, Tong J, Campbell J, D'Alessio DA. High Doses of Exogenous Glucagon Stimulate Insulin Secretion and Reduce Insulin Clearance in Healthy Humans. Diabetes. 2024 Mar 1;73(3):412-425. doi: 10.2337/db23-0201. PMID 38015721
- [Background] Schirra J, Sturm K, Leicht P, Arnold R, Goke B, Katschinski M. Exendin(9-39)amide is an antagonist of glucagon-like peptide-1(7-36)amide in humans. J Clin Invest. 1998 Apr 1;101(7):1421-30. doi: 10.1172/JCI1349. PMID 9525985
- [Background] Salehi M, Aulinger B, Prigeon RL, D'Alessio DA. Effect of endogenous GLP-1 on insulin secretion in type 2 diabetes. Diabetes. 2010 Jun;59(6):1330-7. doi: 10.2337/db09-1253. Epub 2010 Mar 9. PMID 20215429